CLINICAL TRIAL: NCT06693843
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled, Dose-range Finding Study of the Efficacy and Safety of Multiple Doses of Aleniglipron (GSBR-1290) in Participants Living With Obesity (Body Mass Index ≥ 30 kg/m2) or Overweight (Body Mass Index ≥ 27 kg/m2) With at Least One Weight-related Comorbidity
Brief Title: A Phase 2b, Dose-range Finding Study of the Efficacy and Safety of Multiple Doses of Aleniglipron (GSBR-1290) in Participants Living With Obesity or Overweight With at Least One Weight-related Comorbidity
Acronym: ACCESS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gasherbrum Bio, Inc., a wholly owned subsidiary of Structure Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GSBR-1290-06
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Obesity, Overweight, or Chronic Weight Management
Keywords: ACCESS, obesity, overweight, GSBR-1290, aleniglipron, chronic weight management, obese, small molecule, GLP-1 receptor agonist, Structure Therapeutics
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): Participants will receive Aleniglipron or Placebo administered orally.
  Interventions: Drug: Aleniglipron or Placebo
- Cohort 2 (Experimental): Participants will receive Aleniglipron or Placebo administered orally.
  Interventions: Drug: Aleniglipron or Placebo
- Cohort 3 (Experimental): Participants will receive Aleniglipron or Placebo administered orally.
  Interventions: Drug: Aleniglipron or Placebo
- Cohort 1 OLE (Active Comparator): Participants will receive Aleniglipron administered orally
  Interventions: Drug: Aleniglipron
- Cohort 2 OLE (Active Comparator): Participants will receive Aleniglipron administered orally
  Interventions: Drug: Aleniglipron
- Cohort 3 OLE (Active Comparator): Participants will receive Aleniglipron administered orally
  Interventions: Drug: Aleniglipron
- Cohort 4 OLE (Active Comparator): Participants will receive Aleniglipron administered orally
  Interventions: Drug: Aleniglipron

INTERVENTIONS:
Drug: Aleniglipron or Placebo — Drug: Aleniglipron Administered orally Drug: Placebo Administered orally
  Arms: Cohort 1
Drug: Aleniglipron or Placebo — Drug: Aleniglipron Administered orally Drug: Placebo Administered orally
  Arms: Cohort 2
Drug: Aleniglipron or Placebo — Drug: Aleniglipron Administered orally Drug: Placebo Administered orally
  Arms: Cohort 3
Drug: Aleniglipron — Drug: Aleniglipron Administered orally
  Arms: Cohort 1 OLE
Drug: Aleniglipron — Drug: Aleniglipron Administered orally
  Arms: Cohort 2 OLE
Drug: Aleniglipron — Drug: Aleniglipron Administered orally
  Arms: Cohort 3 OLE
Drug: Aleniglipron — Drug: Aleniglipron Administered orally
  Arms: Cohort 4 OLE

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, dose-range finding study of the efficacy, safety, tolerability, PK, and PD of multiple doses of aleniglipron in participants living with overweight or obesity with at least one weight-related comorbidity. Participants will be randomized to aleniglipron or placebo in a ratio of 3:1 within each Cohort receiving multiple-ascending, QD doses of aleniglipron or placebo in titration steps of 4 weeks duration for a total of 36 weeks of treatment. At the end of the study (after completing 36 weeks of treatment), participants will be offered to continue with an open-label extension (OLE) where they will receive aleniglipron for an additional 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* BMI ≥30 kg/m2 or BMI ≥27.0 kg/m2 and previous/current diagnosis of ≥ 1 obesity related comorbidity

Exclusion Criteria:

* Previous documented diagnosis of diabetes mellitus.
* Self-reported change in body weight >5% within 3 months before Screening
* Body weight ≤80 kg at Screening
* Have a prior or planned surgical treatment for obesity (excluding liposuction or abdominoplasty, if performed >1 year prior to screening)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 220 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percent change in body weight from Baseline to Week 36 | Baseline and week 36
  Double Blind Period
TEAEs and SAEs | Baseline and week 72
  Open -Label Extension
AESI | Baseline and week 72
  Open -Label Extension
Evaluate the safety and tolerability of participants with abnormal laboratory values, including hematology, serum chemistry, and coagulation | Baseline and week 72
  Open -Label Extension
Evaluate long-term safety and tolerability of aleniglipron as measured through electrocardiograms (including, but not limited to, the measurements of ventricular HR, PR interval, QRS duration, QT interval, and QTcF) | Baseline and week 72
  Open -Label Extension
Evaluate the safety and tolerability of participants with abnormal vital signs, including blood pressure, heart rate, and temperature | Baseline and week 72
  Open -Label Extension

SECONDARY OUTCOMES:
Percentage of participants who achieve ≥5% reduction in body weight at Week 36 | Baseline and week 36
  Double Blind Period
Percentage of participants who achieve ≥10% reduction in body weight at Week 36 | Baseline and week 36
  Double Blind Period
Percentage of participants who achieve ≥15% reduction in body weight at Week 36 | Baseline and week 36
  Double Blind Period
Change in body weight (absolute) from Baseline to Week 36 | Baseline and week 36
  Double Blind Period
Change in waist circumference from Baseline to Week 36 | Baseline and week 36
  Double Blind Period
Change in body mass index from Baseline to Week 36 | Baseline and week 36
  Double Blind Period
Percent change in body weight | Baseline to week 72 & Week 36-72
  Open -Label Extension
Percentage of participants who achieve ≥5% reduction in body weight | Baseline to week 72 & Week 36-72
  Open -Label Extension
Percentage of participants who achieve ≥10% reduction in body weight | Baseline to week 72 & Week 36-72
  Open -Label Extension
Percentage of participants who achieve ≥15% reduction in body weight | Baseline to week 72 & Week 36-72
  Open -Label Extension
Change in body weight | Baseline to week 72 & Week 36-72
  Open -Label Extension
Change in body mass | Baseline to week 72 & Week 36-72
  Open -Label Extension
Change in waist circumference | Baseline to week 72 & Week 36-72
  Open -Label Extension

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - ACCESS Research Site, Phoenix, Arizona
  - ACCESS Research Site, Anaheim, California
  - ACCESS Research Site, Los Angeles, California
  - ACCESS Research Site, Montclair, California
  - ACCESS Research Site, Rancho Cucamonga, California
  - ACCESS Research Site, Sacramento, California
  - ACCESS Research Site, Spring Valley, California
  - ACCESS Research Site, Honolulu, Hawaii
  - ACCESS Research Site, Chicago, Illinois
  - ACCESS Research Site, Evanston, Illinois
  - ACCESS Research Site, Muncie, Indiana
  - ACCESS Research Site, Valparaiso, Indiana
  - ACCESS Research Site, West Des Moines, Iowa
  - ACCESS Research Site, Baton Rouge, Louisiana
  - ACCESS Research Site, Richfield, Minnesota
  - ACCESS Research Site, City of Saint Peters, Missouri
  - ACCESS Research Site, Hazelwood, Missouri
  - ACCESS Research Site, Springfield, Missouri
  - ACCESS Research Site, Albany, New York
  - ACCESS Research Site, Binghamton, New York
  - ACCESS Research Site, Brooklyn, New York
  - ACCESS Research Site, Rochester, New York
  - ACCESS Research Site, Wilmington, North Carolina
  - ACCESS Research Site, Cincinnati, Ohio
  - ACCESS Research Site, Norman, Oklahoma
  - ACCESS Research Site, Medford, Oregon
  - ACCESS Research Site, Pittsburgh, Pennsylvania
  - ACCESS Research Site, Moncks Corner, South Carolina
  - ACCESS Research Site, Chattanooga, Tennessee
  - ACCESS Research Site, Austin, Texas
  - ACCESS Research Site, Dallas, Texas
  - ACCESS Research Site, Mesquite, Texas
  - ACCESS Research Site, Shavano Park, Texas
  - ACCESS Research Site, West Jordan, Utah
  - ACCESS Research Site, Winchester, Virginia
  - ACCESS Research Site, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address a specific research question in an approved data sharing request
Supporting Information: Study Protocol
Time Frame: Data sharing requests will be considered beginning 36 months after the study publication (manuscript accepted for publication) and either 1) the product has been granted marketing authorization in at least two regulatory jurisdictions, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Researchers will submit a request containing the research objectives, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). Gasherbrum Bio, Inc. does not grant external requests for individual de-identified patient data for the following purposes:
  * re-evaluating safety and efficacy end points already addressed in the product labelling,
  * assessing safety or efficacy for an indication in current development
  Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a panel of external advisors. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement.